CLINICAL TRIAL: NCT00804362
Title: Validation of the Sickle Cell Disease Pain Burden Interview
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, William Zempsky, MD, Director, Pain Relief Program, Connecticut Children's Medical Center
Other Study IDs: 08-093
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Sickle Cell Disease; Pain
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to validate a brief survey tool, the SCD Pain Burden Interview (SCPBI), which can be used in the clinical and/or research settings to assess the impact of pain on children with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Documented sickle cell disease
* 7 years old or greater
* Primary caregiver present at the first visit for children < 18 years of age

Exclusion Criteria:

* Primary language spoken other than English
* Patient is in acute pain episode at time of initial visit

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents diagnosed with sickle cell disease.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Correlation with validated measures of pain interference, function, quality of life, and mood. | Quarterly

CONTACTS AND LOCATIONS:
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States